CLINICAL TRIAL: NCT01756469
Title: Alcohol Harm Reduction Intervention Among Female Sex Workers in Mombasa, Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PHE#KE.09.0235
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Alcohol Use and STI/HIV Infections, Domestic Violence
MeSH Terms: conditions — Alcohol Drinking | interventions — Behavior Therapy; Ethanol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): non-alcohol related information about nutrition
- Intervention (Active Comparator): Behavioral Intervention for Alcohol Use
  Interventions: Behavioral: Behavioral Intervention for Alcohol Use

INTERVENTIONS:
Behavioral: Behavioral Intervention for Alcohol Use — Behavioral Intervention for Alcohol Use
  Other Names: BI
  Arms: Intervention

SUMMARY:
The main study objective is to investigate whether female sex workers (FSWs) at drop-in centers in Mombasa, Kenya, who report harmful or hazardous alcohol intake and participate in a brief alcohol intervention (vs. those who participate in a nutrition intervention in the control group), will reduce their alcohol use and incidence of STIs, HIV, and sexual violence, as well as increase their condom use.

DETAILED DESCRIPTION:
This is a longitudinal intervention study among female sex workers affiliated with the APHIA II program, who have harmful or hazardous alcohol use patterns. The purpose of the study is to obtain initial estimates of the impact of the intervention on alcohol use and STI acquisition, to help determine if this is a program that should be implemented more fully. Female sex workers will be recruited from three APHIA drop-in centers in Mombasa district, Kenya who serve more than 15,000 FSWs. Approximately 800 FSWs with harmful or hazardous alcohol use will be enrolled in the study over a six-month accrual period with a follow-up of 12 months for each participant. FSWs will be randomly assigned to either the intervention or "active" control arm. The intervention arm will receive the Brief Intervention for Alcohol Use (BI), which is designed for individuals with harmful or hazardous alcohol use, in addition to information about nutrition. The control arm will receive only non-alcohol related information about nutrition during the study period. A peer educator from the APHIA II project will inform potential participants about the study. A trained nurse counselor or research assistant will then screen interested volunteers for harmful alcohol use with the validated AUDIT questionnaire (WHO, 2001) and obtain informed consent from eligible participants. Arm assignment using random allocation will be made after volunteers are screened for eligibility, provide consent for participation, and complete baseline data collection procedures. Follow-up data collection will occur at six and twelve months post-randomization. Data collection procedures at all three time points will include the AUDIT questionnaire, a behavioral interview, a gynecological exam including STI diagnosis and treatment, and a HIV rapid test and counseling.

ELIGIBILITY:
Inclusion Criteria:

* Female sex worker, defined as a woman who self reports exchange of any type of sex including oral, anal, and vaginal sex for money or gifts within the six months prior to study enrollment;
* Self-identifies as a woman;
* 18 years or older;
* Scores between 7-19 on the AUDIT questionnaire;
* Willing to participate in the study and all data collection procedures;
* Lives in Mombasa or plans on residing in Mombasa for 12 months following study enrollment;
* Currently participating in the APHIA II sex worker peer education program; and
* Documentation of negative tests for gonorrhea, Chlamydia, and trichomoniasis.

Exclusion Criteria:

* Scores less than 7 (low-risk drinking) or more than 19 (high-risk drinking/alcohol dependence) on the AUDIT questionnaire;
* Plans to be away in the next 12 months for more than six months or relocate away from the study site;
* Currently participating in another HIV intervention study; or
* Has any other condition that, in the opinion of the investigator or designee, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise with achieving the study objectives.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 818 (Actual)
Dates: Start 2011-03; Primary Completion 2012-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Alcohol use and STI/HIV infection | up to 12 months
  Outcomes assessed at up to 12 months follow-ups

SECONDARY OUTCOMES:
Condom use and sexual violence | up to 12 months
  Outcomes assessed at up to 12 months follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Peter Mwarogo, MPH, Principal Investigator — FHI 360
Locations (1):
- FHI360, Nairobi, Kenya

REFERENCES:
- [Derived] Greene MC, Kane J, Alto M, Giusto A, Lovero K, Stockton M, McClendon J, Nicholson T, Wainberg ML, Johnson RM, Tol WA. Psychosocial and pharmacologic interventions to reduce harmful alcohol use in low- and middle-income countries. Cochrane Database Syst Rev. 2023 May 9;5(5):CD013350. doi: 10.1002/14651858.CD013350.pub2. PMID 37158538